CLINICAL TRIAL: NCT03406858
Title: Phase II Trial of Immune Checkpoint Inhibitor With Anti-CD3 x Anti-HER2 Bispecific Antibody Armed Activated T Cells in Metastatic Castrate Resistant Prostate Cancer
Brief Title: Pembro and HER2Bi-Armed Activated T Cells in Treating Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abhinav Deol, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-135; NCI-2017-02156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-135 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2018-01-23 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Prostate Carcinoma Metastatic in the Bone; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, HER2Bi-armed activated T cells) (Experimental): Patients receive pembrolizumab IV over 30 minutes every 3 weeks. Treatment repeats every 3 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity. Beginning at least 1 week after pembrolizumab, patients receive HER2Bi-armed activated T cells IV over 5-15 minutes 2 times a week for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: HER2Bi-Armed Activated T Cells; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Biological: HER2Bi-Armed Activated T Cells — Given IV
  Other Names: Anti-CD3 x Anti-Her2/neu Bispecific Antibody-Armed Activated T Cells; HER2Bi-Armed ATCs
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and HER2Bi-armed activated T cells work in treating patients with castration resistant prostate cancer that has spread to other places in the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. HER2Bi-armed activated T cells are made using T cells and may target and kill cancer cells. Giving pembrolizumab and HER2Bi-armed activated T cells may work better in treating patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical efficacy of 8 infusions of HER2 HER2Bi-armed activated T cells (BATs) (up to 10^10/infusion) twice per week for 4 weeks in combination with pembrolizumab once every 3 weeks starting with one dose 3 weeks before the 1st BATs infusion, by assessing the percentage of patients free of clinical progression at 6 months after registration.

SECONDARY OBJECTIVES:

I. Evaluate phenotype, cytokine profiles and IFN-gamma enzyme-linked immunosorbent spots (ELISpots), cytotoxicity and antibodies directed at laboratory prostate cancer cell lines for proof of principle of immune system activation and to correlate with clinical outcomes of response, progression free survival (PFS), and overall survival (OS).

II. Evaluate the magnitude of change in tumor infiltrating T cells, PD-1 expression, and the Th1/Th2 ratio in prostate cancer tumor tissue before and after immunotherapy and correlate it with the clinical outcomes of response, PFS, and OS.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes every 3 weeks. Treatment repeats every 3 weeks for up to 6 months in the absence of disease progression or unacceptable toxicity. Beginning at least 1 week after pembrolizumab, patients receive HER2Bi-armed activated T cells IV over 5-15 minutes 2 times a week for 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have histologically confirmed prostate adenocarcinoma, with metastases
* Progression by either PSA, Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria for measurable disease or new areas of metastases on bone scan or symptom progression related to prostate cancer despite castrate levels of testosterone; (level < 50 ng/ml)
* Be agreeable to continue to maintain castrate levels of testosterone
* At least 2 weeks should have elapsed since any immunosuppressive therapy
* At least 4 weeks since prior chemotherapy for metastatic disease or at least 2 weeks since prior androgen targeting agents such as ketoconazole, abiraterone, enzalutamide, etc.
* Discontinue anti-androgens prior to therapy; at least 6 weeks since last dose of bicalutamide or nilutamide and at least 4 weeks from last dose of flutamide
* Have normal bone marrow, renal and hepatic function as deemed by the treating physician and approved by the clinical principal investigator (PI) Dr. Vaishampayan
* Not have concurrent anti-cancer therapy
* Not have concurrent immunosuppressive therapy or medical condition likely to cause immunosuppression
* Have life expectancy > 6 months
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG)/Zubrod performance scale
* Agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Within 10 days of treatment registration: Absolute neutrophil count (ANC) >= 1,500 /mcL
* Within 10 days of treatment registration: Platelets >= 100,000 / mcL
* Within 10 days of treatment registration: Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Within 10 days of treatment registration: Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Within 10 days of treatment registration: Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Within 10 days of treatment registration: Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT] =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Within 10 days of treatment registration: Albumin >= 2.5 mg/dL
* Within 10 days of treatment registration: International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Within 10 days of treatment registration: Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg of prednisone daily or equivalent steroid doses) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Has hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or has not recovered (i.e. =< grade 1 or at baseline) from adverse events due to agents administered earlier; Note: Subjects with =<grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Has received major surgery, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g. hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g. hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated vaccines, and are not allowed
* Has history of cardiac or pulmonary impairment either by clinical history or symptoms or cardiac ejection fraction < 40%

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Deol, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient went through Pheresis but did not return for treatment. They were excluded from the Progression-Free Survival analysis but were included in adverse events since they began the process.
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells)
Started | 15
Completed | 13
Not Completed | 2
Not completed — Failure to receive treatment drug. | 1
Not completed — ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 69 [57 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Percentage of patients achieving clinical progression-free interval at 6 months from study registration
Time Frame: Up to 6 months
Population: All patients that received treatment. One patient went through Pheresis but never returned for treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells)
Number analyzed (Participants) | 13
percentage of participants | 38.5 [19.3 to 76.5]

ADVERSE EVENTS:
Time Frame: For the time period beginning at treatment allocation/randomization through 90 days following cessation of treatment, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier, up to 6 months.
Arm/Group | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells)
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells) (N=14)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, HER2Bi-armed Activated T Cells) (N=14)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Chills (General disorders) | 9 (9)
Cholesterol high (Investigations) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 11 (12)
Fever (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (6)
Headache (Nervous system disorders) | 7 (7)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Edema limbs (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to COVID-19 pandemic, cellular therapies were suspended and hence the study was discontinued before the targeted enrollment was reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT03406858/Prot_SAP_000.pdf